CLINICAL TRIAL: NCT04210505
Title: Povidone-iodine to Stop Access-related Infections and Transmission of Staphylococcus Aureus (PAINTS)
Brief Title: Nasal Decolonization of Dialysis Patients Noses
Acronym: PAINTS
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Marin L. Schweizer, PhD (Other)
Collaborators: University of Pennsylvania (Other); University of Illinois at Chicago (Other); Washington University School of Medicine (Other); Emory Healthcare (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); 3M (Industry)
Responsible Party: Sponsor-Investigator, Marin L. Schweizer, PhD, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pending; 1R01HS026724 (AHRQ)
Record Dates: First submitted 2019-12-18; First posted 2019-12-24 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Staphylococcus Aureus Infection
Keywords: Dialysis; povidone-iodine
MeSH Terms: conditions — Staphylococcal Infections | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nasal Povidone-Iodine Decolonization Intervention (Experimental): Intranasal povidone-iodine (3M Skin and Nasal Antiseptic) will be applied to the patients' noses at each hemodialysis session.
  Interventions: Drug: Povidone-Iodine Topical Ointment; Other: Standard Care
- Concurrent Control (No Intervention): Standard of Care. This will be usual care at each hemodialysis center.

INTERVENTIONS:
Drug: Povidone-Iodine Topical Ointment — Intranasal povidone-iodine will be applied to the lower anterior nares (i.e. nostril) of patients undergoing hemodialysis before each session.
  Arms: Nasal Povidone-Iodine Decolonization Intervention
Other: Standard Care — Control group will receive standard care as provided by the dialysis center
  Arms: Nasal Povidone-Iodine Decolonization Intervention

SUMMARY:
Hemodialysis patients are at high-risk for infections, specifically Staphylococcus aureus infections. The investigators propose to 1) implement a novel intervention (nasal povidone-iodine at each hemodialysis session) to prevent S. aureus infections using a stepped-wedge cluster randomized trial, and 2) evaluate the feasibility and acceptability of this intervention. If successful, this intervention can be used among hemodialysis patients, and evaluated in other high-risk patient populations to prevent S. aureus infections.

DETAILED DESCRIPTION:
The PAINTS study is a stepped-wedge cluster randomized trial that will compare standard care to an intervention that includes nasal povidone-iodine at each hemodialysis session to determine whether nasal povidone-iodine prevents infections. The nasal povidone-iodine will be donated by 3M. This formulation of nasal povidone-iodine was developed under the Tentative Final Monograph for Health-Care Antiseptic Drug Products 21 CFR Parts 333 and 369 (Docket # 75N-183H), Federal Register Volume 59, Number 116, Friday, June 17, 1994, Proposed Rules. However, the product need not be controlled like a pharmaceutical drug. The product may be stored and controlled similarly to an iodine or alcohol skin preparation product.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients receiving outpatient chronic hemodialysis at one of the 16 study dialysis centers.

Note: the unit of randomization is the dialysis center, not the individual patient

Exclusion Criteria:

Patients receiving peritoneal dialysis or home hemodialysis Pregnant women Patients with known sensitivity or allergy to iodine (documented or verbalized) Patients with active bacterial infections Children < 18 years of age. Patients with infections at the beginning of the study will enter the study after antibiotic treatment is complete.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Staphylococcus aureus bloodstream infection | Through study completion (up to 3 years)
  Centers for Disease Control and Prevention (CDC) National Healthcare Safety Network (NHSN) definition: a Staphylococcus aureus positive blood specimen collected in the outpatient setting or within 1 calendar day after a hospital admission

SECONDARY OUTCOMES:
Incidence of Staphylococcus aureus access related bloodstream infection (ARBSI) | Through study completion (up to 3 years)
  Centers for Disease Control and Prevention (CDC) National Healthcare Safety Network (NHSN) definition: a Staphylococcus aureus bloodstream infection with the suspected source reported as the vascular access or uncertain
Incidence of Staphylococcus aureus local access site infection | Through study completion (up to 3 years)
  Centers for Disease Control and Prevention (CDC) National Healthcare Safety Network (NHSN) definition: pus, redness or increased swelling at the vascular access site when an ARBSI is not present but with positive culture for Staphylococcus aureus
Incidence of Bloodstream infections by any pathogen | Through study completion (up to 3 years)
  Centers for Disease Control and Prevention (CDC) National Healthcare Safety Network definition: a positive blood specimen collected in the outpatient setting or within 1 calendar day after a hospital admission
Incidence of Access related bloodstream infection by any pathogen | Through study completion (up to 3 years)
  Centers for Disease Control and Prevention (CDC) National Healthcare Safety Network definition: a bloodstream infection with the suspected source reported as the vascular access or uncertain
Incidence of Local access site infection | Through study completion (up to 3 years)
  Centers for Disease Control and Prevention (CDC) National Healthcare Safety Network (NHSN) definition: pus, redness or increased swelling at the vascular access site when an ARBSI is not present
Incidence of Staphylococcus aureus bloodstream infection among patients who agreed to participate in intervention | Through study completion (up to 3 years)
  Centers for Disease Control and Prevention (CDC) National Healthcare Safety Network

CONTACTS AND LOCATIONS:
Overall Officials: Marin L Schweizer, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (5):
- United States (5):
  - Emory Healthcare, Atlanta, Georgia
  - University of Illinois Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Washington University, St Louis, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The investigators will submit an electronic version of each peer-reviewed accepted manuscript to PubMed Central to be made publicly available within 12 months of publication. The investigators will respond to requests for restricted public health data sets and ensure responses follow appropriate processes, documentation, and approval.
Supporting Information: Study Protocol
Time Frame: Until year 2025
Access Criteria: Upon request

REFERENCES:
- [Derived] Armstrong-Pavlik F, Racila AM, Ward M, Nair R, Tolomeo P, Kellogg J, Lindsey B, Herwaldt LA, Jacob JT, Vijayan A, Pegues D, Cobb J, Fraer M, Casey SB, Dukes KC, Hockett Sherlock S, Hopps M, Schweizer ML. Survey of hemodialysis patients' knowledge of their infection risk and acceptability of an intranasal decolonization intervention. Infect Control Hosp Epidemiol. 2026 Feb 4:1-5. doi: 10.1017/ice.2025.10386. Online ahead of print. PMID 41635193
- [Derived] Racila AM, O'Shea AMJ, Nair R, Dukes K, Herwaldt LA, Boyken L, Diekema D, Ward MA, Cobb J, Jacob J, Pegues D, Bleasdale S, Vijayan A, Mutneja A, Fraer M, O'Connell-Moore D, Tolomeo P, Mendez M, Jaworski E, Schweizer ML. Using nasal povidone-iodine to prevent bloodstream infections and transmission of Staphylococcus aureus among haemodialysis patients: a stepped-wedge cluster randomised control trial protocol. BMJ Open. 2021 Dec 3;11(12):e048830. doi: 10.1136/bmjopen-2021-048830. PMID 34862278

DOCUMENTS (1):
  • Informed Consent Form (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/05/NCT04210505/ICF_000.pdf